CLINICAL TRIAL: NCT03247608
Title: ConnectedHeartHealth - Heart Failure Readmission Intervention
Acronym: CHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: American Heart Association (AHA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB #2287; CHH (Other: LifeBridge Health)
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease; Heart Failure
Keywords: Ambio Health
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ambio Health Remote Monitoring (Experimental): Ambio Health is an end-to-end remote patient monitoring system which includes a weight scale, blood pressure meter and blood glucose meter with wireless transmission of biometric readings through a home gateway to a web-based care management application that provides population health remote patient monitoring and engagement with automated delivery of the CarePlans.
  Interventions: Behavioral: Ambio Health Remote Monitoring

INTERVENTIONS:
Behavioral: Ambio Health Remote Monitoring — Participants in the Connected Heart Health study will complete a 24 week CarePlan including education, biometric monitoring, and communication with the health care team members. Each day the participant will receive an email from Ambio Health with a daily task list that includes a variety of activities. These tasks include uploading biometrics (weight and blood pressure), completing assessment on self-management skills (nutrition, physical activity, and medication management), accessing educational content (videos, web links, interactive quizzes), participation in challenges, and communicating with the care team and care givers.

SUMMARY:
This is a single-center, pilot study that will evaluate the effectiveness of the AHA science based CarePlans and the Ambio Health technology in improving the risk adjusted 30 day readmissions rate, patient compliance, and biometrics. The study will also be used to assess the feasibility of similar heart failure transition programs in the future.

DETAILED DESCRIPTION:
A key strategy of the Affordable Care Act is the Accountable Care Organization, designed to improve the quality of care, promote population health and reduce costs by making healthcare providers more accountable for health outcomes. With the increasing pressure to simultaneously improve care and reduce the overall cost of care, there is increasing need for better care coordination, especially for patients that are high risk for readmissions and poor health outcomes, to stay connected with their healthcare provider outside of the healthcare setting. Connected Heart Health is the American Heart Association's ACO (Accountable Care Organization) strategy for post-acute care. This includes evidence based CarePlans for heart failure, cardiac rehabilitation, and coronary artery disease. These CarePlans are brought to life with technology enabled by Ambio Health, which allows patients and doctors to be connected anytime and anywhere, encouraging the adoption of self-management skills, healthy living, and evidence based practice, resulting in fewer cardiovascular events and readmissions, and lower costs.

Ambio Health is an end-to-end remote patient monitoring system which includes a weight scale, blood pressure meter and blood glucose meter with wireless transmission of biometric readings through a home gateway to a web-based care management application that provides population health remote patient monitoring and engagement with automated delivery of the CarePlans.

Ambio Health will be introduced as a viable method for remote monitoring of heart failure patients, with an emphasis on reducing readmission rates and promoting self-management skills. This program is intended to implement the AHA's Connected Heart Health CarePlan and educational content for patients in conjunction with a platform designed to upload biometric data and provide care coordination as directed and implemented by discharging physicians/institutions. The intent is to design and execute a Pilot with Sinai Hospital of Baltimore.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Heart Failure as measured by the New York Heart Association (NYHA) functional classification and is currently in functional class II- IV status.
* Have been hospitalized for an episode of acute HF decompensation within the last 30 days.
* Have access to the internet.
* Are physically and mentally capable to complete the monitoring process or have a caregiver capable of assisting in the use of the Ambio Health system.
* Willing and able to sign an informed consent form to participate in this evaluation for a duration of 180 days.

Exclusion Criteria:

* Have a life expectancy of less than six months.
* Live in a nursing home other multi-member assisted living facility
* Intend to be away from their home for more than 2 weeks (14 days) total during the monitoring period.
* Are unable to read English at a minimum 5th grade level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Re-admissions rate | 30 Days
  The primary endpoint will be the risk adjusted 30 day readmissions rate of the study population in comparison with the Sinai Hospital and the National Average.

SECONDARY OUTCOMES:
Compliance to guidelines measures | 30 Days
  Additional study metrics will include compliance to evidence based guidelines using Get with the Guidelines HF measures.
Biometrics change | 30 Days
  Additional study metrics will include change in biometrics from baseline to follow up for weight, blood pressure and pro-BNP.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Moscucci, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No